CLINICAL TRIAL: NCT04755712
Title: Comparison of Two Analgesic Strategies After Scheduled Caesarean : Block of the Lumbar Region With Ropivacaine Versus Intrathecal Morphine
Brief Title: Comparison of Two Analgesic Strategies After Scheduled Caesarean
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-A03334-35
Record Dates: First submitted 2021-02-08; First posted 2021-02-16 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2022-10

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine; Sufentanil; Sodium Chloride; Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ropivacaine in quadratum lumburum block 2 (Experimental): Ropivacaine will be administrated in perineural in quadratum lumburum block 2 after the caesarian.
  Interventions: Drug: Rachianesthesia; Drug: Morphine
- Intrathecal morphine (Active Comparator): Morphine will be administrated in intrathecal
  Interventions: Drug: Rachianesthesia; Drug: Sodium Chloride Injection; Drug: Morphine

INTERVENTIONS:
Drug: Rachianesthesia — Administration of different anesthesia drugs in accordance with the courant practice (mixture of bupivacaine and sufentanil)
  Other Names: Bupivacaine and sufentanil
Drug: Sodium Chloride Injection — Subcutaneous injection of Sodium chloride at the usual quadratum lumburum block 2 (QLB2) injection site under ultrasound ("sham-QLB2").
  Other Names: sham-QLB2
  Arms: Intrathecal morphine
Drug: Morphine — Morphine via pump (patient controlled analgesia)
  Other Names: injection of morphine

SUMMARY:
To demonstrate the superiority of square lumbar block to ropivacaine compared to intrathecal morphine in the efficacy of postoperative analgesia following scheduled caesarean.

DETAILED DESCRIPTION:
Interventional, comparative, randomized, controlled study versus reference therapeutic strategy, in 2 parallel groups, double-blind (patient and evaluator), single-center, aiming to demonstrate the superiority of ropivacaine in square lumbar block versus intrathecal morphine, on the efficacy of post-operative analgesia, following a scheduled caesarean.

ELIGIBILITY:
Inclusion Criteria:

* Patient to undergo a scheduled caesarean under spinal anesthesia, for the birth of a term baby with a Pfannenstiel-type incision;
* Patient in good health ;
* Patient able to understand the information related to the study, read the information leaflet and agree to sign the consent form.

Exclusion Criteria:

* Pregnancy less than 37 weeks with amenorrhea;
* Multiple pregnancy;
* Fetal pathology known at the time of inclusion;
* Body mass index> 45 kg / m²;
* History of scoliosis or spine surgery;
* History of chronic pain associated with taking opiates, neuropathic pain, neurological pathology;
* Preoperative anemia (blood hemoglobin <9 g / dL);
* Hypersensitivity to ropivacaine or other local anesthetics with amide bond;
* Hypersensitivity to morphine or opioids;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Cumulative quantity of morphine received postoperatively via pump | 1 day
  The main objective of the study is to demonstrate the superiority of square lumbar block to ropivacaine (quadratum lumburum block 2 - QLB2) in comparison to intrathecal morphine in the efficacy of postoperative analgesia following a scheduled Caesarean.

SECONDARY OUTCOMES:
Characteristics of postoperative pain using a visual analogic scale | 2 days
  Evaluate the characteristics of postoperative pain in both groups with the use of a visual analog scale
Side effects of the two analgesic strategies | 2 days
  Evaluate the side effects of the two analgesic strategies reported in a case report form
Cumulative quantity of morphine received postoperatively via pump | 2 days
  Demonstrate the superiority of square lumbar block to ropivacaine (quadratum lumburum block 2 - QLB2) in comparison to intrathecal morphine in the efficacy of postoperative analgesia following a scheduled Caesarean.

CONTACTS AND LOCATIONS:
Locations (1):
- MAUPAIN, Quincy-sous-Sénart, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giral T, Delvaux BV, Huynh D, Morel B, Zanoun N, Ehooman F, Garnier T, Maupain O. Posterior quadratus lumborum block versus intrathecal morphine analgesia after scheduled cesarean section: a prospective, randomized, controlled study. Reg Anesth Pain Med. 2026 Jan 5;51(1):82-89. doi: 10.1136/rapm-2024-105454. PMID 39237149